CLINICAL TRIAL: NCT04915339
Title: Pilot Study Among Type 2 Diabetes Patients Investigating Effects of Computerized Cognitive and Physical Activity Programs Combined or Single.
Brief Title: Pilot Study Among Type 2 Diabetes Patients Investigating the Effects of Computerized Cognitive and Physical Activity Programs Combined or Single (DIASCOP)
Acronym: DIASCOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University of Clermont Auvergne (UCA) / LAPSCO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: RBHP 2020 DUTHEIL; 2020-A03228-31 (Other: ANSM)
Record Dates: First submitted 2021-05-21; First posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Physical fitness; Neuropsychological Tests; Cognition; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise; Cognitive Training

STUDY DESIGN:
Intervention Model Description: * Group 1: physical activity (one month) then cognitive training (one month)
  * Group 2: Cognitive training (one month) then physical activity (one month)
  * Group 3 : resonance frequency breathing (one month) then combined physical activity and cognitive (one month) training
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study hypothesis is not given to the participants and the investigator will not be aware of the group the participants have been allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: physical activity then cognitive training (Experimental): Using an online-computerized application, physical activities will be prescribed for one month. After a 15 days break, cognitive training activities will be prescribed the same way. A feedback by the patient will be asked fallowing each activity to control the observance.
  Interventions: Behavioral: Physical activity; Behavioral: cognitive training
- Group 2: Cognitive training then physical activity (Experimental): Contrary to the first group, the second one starts with cognitive training intervention then engages in physical activity in same way as the first group. A feedback by the patient will also be asked fallowing each activity to control the observance
  Interventions: Behavioral: Physical activity; Behavioral: cognitive training
- Group 3 : resonance frequency breathing then combined physical activity and cognitive training (Experimental): The third group takes part in a 1 month breathing exercise program. After a 15 days break (as the groups 1 and 2), a combined physical activity and cognitive training program is administrated for 1 month. As the others arms, a feedback by the patient will be asked fallowing each activity to control the observance
  Interventions: Behavioral: combined physical and cognitive training

INTERVENTIONS:
Behavioral: Physical activity — The intervention is administrated through a computerized application as prescribed exercises (cognitive or physical). The specific measures that will be used to determine the effect of the intervention are psychological variables (mood, anxiety, well-being, cognitive variables…) and physical ones (Heart rate variability, stress biomarkers, fat and muscle mass, blood circulation…).
  Arms: Group 1: physical activity then cognitive training; Group 2: Cognitive training then physical activity
Behavioral: cognitive training — The intervention is administrated through a computerized application as prescribed exercises (cognitive or physical). The specific measures that will be used to determine the effect of the intervention are psychological variables (mood, anxiety, well-being, cognitive variables…) and physical ones (Heart rate variability, stress biomarkers, fat and muscle mass, blood circulation…).
  Arms: Group 1: physical activity then cognitive training; Group 2: Cognitive training then physical activity
Behavioral: combined physical and cognitive training — The intervention is administrated through a computerized application as prescribed exercises (cognitive or physical). The specific measures that will be used to determine the effect of the intervention are psychological variables (mood, anxiety, well-being, cognitive variables…) and physical ones (Heart rate variability, stress biomarkers, fat and muscle mass, blood circulation…).
  Arms: Group 3 : resonance frequency breathing then combined physical activity and cognitive training

SUMMARY:
The purpose of this study is to assess the cognitive benefits of combined physical activity and cognitive training on cognitive health compare to physical activity or cognitive training programs singly administrated among type 2 diabetes. Two group in cross over will take part in either physical activity only (for the first one) or cognitive training only (for the second one) for one month then the other way around during the second month. A fallow up will be administrated 3 months later.

DETAILED DESCRIPTION:
The growing Type 2 diabetes prevalence is associated with health, economic and social consequences. As such, type 2 diabetes is recognized as major health issue. Health care should go on after being discharged from the hospital in order to promote cognitive autonomy. Physical activity and cognitive training are two interventions often recommended individually to benefit cognition among type 2 diabetes patients. Yet, a program combining physical activity and cognitive training might be more effective to favor cognitive health.

In this study, diabetes patient between 50 and 75 years old will be allocated randomly in 3 intervention groups in order to have a homogeneous distribution of the education level, sex and age across the 3 samples. The first group will take part in a physical activity program the first month and in a cognitive training one the second. The second group will be cross-over meaning taking part in a cognitive training program the first month and engaging in the physical activity one the second month. The last group will engage in a program based on resonance frequency breathing the first month (as a control condition), then in a combined physical activity and cognitive training program. Between the 2 interventions, there will be a 15 days break (limiting the transfer of the effect of one intervention onto another). At the beginning of the study, a screening will allow to identify possible exclusion criteria (health factors that could influence the main outcomes). At the beginning (baseline) of the first intervention and after each month, neuropsychological tests assessing cognitive and psychological health as well as well-being. Physiological parameters such as heart rate variability, cortisol and DHEA levels, muscle and lean mass, blood circulation (assessed by Laser speckle contrast imaging). A whole session (psychological and physiological testing) should take 1 h 30. Besides, participants will complete online questionnaires. They have one week after the testing to complete those surveys. If they are late an email will be sent before a phone call in the case the delay goes on.

The main outcome is the increase of the cognitive variables after the intervention. It is expected that the physical activity and cognitive training combined program will benefit cognitive functioning more than either of those programs administrated individually. To investigate to long-term effects of the intervention, a fallow up 3 months later will be conduct

ELIGIBILITY:
Inclusion Criteria:

Male or female aged between 50 and 70 years old, suffering from type 2 diabetes.

Normal or corrected sight and audition. Being able to engage in physical activity. Being able to give enlightened consent. Being affiliate to social welfare

Exclusion Criteria:

Being unable to meet the study conditions or to answer in French to surveys. Any condition considered, by the investigator, as incompatible with the participation in the study.

Major incapacities. Refusal of participation.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Episodic memory performances | Month 1 (Between 1 day and a week before and after the first intervention)
  Scores are obtained from delayed memory recall tests from the logical memory subtest of the Wechsler memory scale. It consists of two short narrative stories with an immediate recall phase after each story and a delayed recall phase after 10 minutes. During the delayed recall, each correct detail was awarded with one score point. On a scale of 0 to 50, a higher score means a better detailed recall.
Episodic memory performances | Month 2 (a week after the second intervention)
  Scores are obtained from delayed memory recall tests from the logical memory subtest of the Wechsler memory scale. It consists of two short narrative stories with an immediate recall phase after each story and a delayed recall phase after 10 minutes. During the delayed recall, each correct detail was awarded with one score point. On a scale of 0 to 50, a higher score means a better detailed recall.
Episodic memory performances | Month 3
  Scores are obtained from delayed memory recall tests from the logical memory subtest of the Wechsler memory scale. It consists of two short narrative stories with an immediate recall phase after each story and a delayed recall phase after 10 minutes. During the delayed recall, each correct detail was awarded with one score point. On a scale of 0 to 50, a higher score means a better detailed recall.

SECONDARY OUTCOMES:
Heart rate variability | Month 1 (Between 1 day and a week before and after the first intervention)
  Time interval between two heart beats assessed by a monitoring watch (Empatica E4) and belt (Zephyr Bioharness 3)
Heart rate variability | Month 2 (a week after the second intervention)
  Time interval between two heart beats assessed by a monitoring watch (Empatica E4) and belt (Zephyr Bioharness 3)
Heart rate variability | Month 3
  Time interval between two heart beats assessed by a monitoring watch (Empatica E4) and belt (Zephyr Bioharness 3)
Blood circulation | Month 1 (Between 1 day and a week before and after the first intervention)
  Assessed by laser speckle contrast imaging (LSCI).
Blood circulation | Month 2 (a week after the second intervention)
  Assessed by laser speckle contrast imaging (LSCI).
Blood circulation | Month 3
  Assessed by laser speckle contrast imaging (LSCI).
Biomarkers of stress | Month 1 (Between 1 day and a week before and after the first intervention)
  A salivary sample to test cortisol level and DHEA.
Biomarkers of stress | Month 2 (a week after the second intervention)
  A salivary sample to test cortisol level and DHEA.
Biomarkers of stress | Month 3
  A salivary sample to test cortisol level and DHEA.
Body Mass index | Month 1 (Between 1 day and a week before and after the first intervention)
  The ratio between weight and height will be computed to report BMI in kg/m2.
Body Mass index | Month 2 (a week after the second intervention)
  The ratio between weight and height will be computed to report BMI in kg/m2.
Body Mass index | Month 3
  The ratio between weight and height will be computed to report BMI in kg/m2.
Life satisfaction scale | Month 1 (Between 1 day and a week before and after the first intervention)
  This scale assesses the feeling of satisfaction of one's life. This scale has 5 items. The minimum score is 5 and the maximum score is 35. A higher score means a higher life satisfaction level.
Life satisfaction scale | Month 2 (a week after the second intervention)
  This scale assesses the feeling of satisfaction of one's life. This scale has 5 items. The minimum score is 5 and the maximum score is 35. A higher score means a higher life satisfaction level.
Life satisfaction scale | Month 3
  This scale assesses the feeling of satisfaction of one's life. This scale has 5 items. The minimum score is 5 and the maximum score is 35. A higher score means a higher life satisfaction level.
Psychological Outcome Profiles | Month 1 (Between 1 day and a week before and after the first intervention)
  This survey assesses the patient's satisfaction level before and after the intervention. Five items with a 6-points Likert scale (0 to 5) allow to obtain a score between 0 and 25. A higher score means a better satisfaction level
Psychological Outcome Profiles | Month 2 (a week after the second intervention)
  This survey assesses the patient's satisfaction level before and after the intervention. Five items with a 6-points Likert scale (0 to 5) allow to obtain a score between 0 and 25. A higher score means a better satisfaction level
Psychological Outcome Profiles | Month 3
  This survey assesses the patient's satisfaction level before and after the intervention. Five items with a 6-points Likert scale (0 to 5) allow to obtain a score between 0 and 25. A higher score means a better satisfaction level
Interoception awareness questionnaire | Month 1 (Between 1 day and a week before and after the first intervention)
  To assess the awareness of both neutral and negative bodily signals, this scale has 19 items with a 5-points Likert scale (1 to 5). The minimum total score is 9 while the maximum is 95. A higher score means a higher perception of bodily signals.
Interoception awareness questionnaire | Month 2 (a week after the second intervention)
  To assess the awareness of both neutral and negative bodily signals, this scale has 19 items with a 5-points Likert scale (1 to 5). The minimum total score is 9 while the maximum is 95. A higher score means a higher perception of bodily signals.
Interoception awareness questionnaire | Month 3
  To assess the awareness of both neutral and negative bodily signals, this scale has 19 items with a 5-points Likert scale (1 to 5). The minimum total score is 9 while the maximum is 95. A higher score means a higher perception of bodily signals.
BORB Birmingham Object Recognition Battery | Month 1 (Between 1 day and a week before and after the first intervention)
  To assess visuospatial processing by asking the participants if two stimuli are orientated the same way.
BORB Birmingham Object Recognition Battery | Month 2 (a week after the second intervention)
  To assess visuospatial processing by asking the participants if two stimuli are orientated the same way.
BORB Birmingham Object Recognition Battery | Month 3
  To assess visuospatial processing by asking the participants if two stimuli are orientated the same way.
Executive functions | Month 1 (Between 1 day and a week before and after the first intervention)
  A battery of 5 tests assessing cognitive inhibition (Stroop and Go/No-Go), cognitive flexibility (Trail Making Test), working memory (Nback) and lexical access (verbal fluency) to reflect executive functioning.
Executive functions | Month 2 (a week after the second intervention)
  A battery of 5 tests assessing cognitive inhibition (Stroop and Go/No-Go), cognitive flexibility (Trail Making Test), working memory (Nback) and lexical access (verbal fluency) to reflect executive functioning.
Executive functions | Month 3
  A battery of 5 tests assessing cognitive inhibition (Stroop and Go/No-Go), cognitive flexibility (Trail Making Test), working memory (Nback) and lexical access (verbal fluency) to reflect executive functioning.
The emotion regulation questionnaire | Month 1 (Between 1 day and a week before and after the first intervention)
  A questionnaire to measure emotion regulation strategies one favors such as emotion suppression or cognitive reappraisal. This questionnaire has 10 items with a 5-points Likert scale (1 to 5). The score ranges from 5 to 50. A higher score means better emotion regulation strategies.
The emotion regulation questionnaire | Month 2 (a week after the second intervention)
  A questionnaire to measure emotion regulation strategies one favors such as A questionnaire to measure emotion regulation strategies one favors such as emotion suppression or cognitive reappraisal. This questionnaire has 10 items with a 5-points Likert scale (1 to 5). The score ranges from 5 to 50. A higher score means better emotion regulation strategies.
The emotion regulation questionnaire | Month 3
  A questionnaire to measure emotion regulation strategies one favors such as emotion suppression or cognitive reappraisal. This questionnaire has 10 items with a 5-points Likert scale (1 to 5). The score ranges from 5 to 50. A higher score means better emotion regulation strategies.
Beck Depression Scale | Month 1 (Between 1 day and a week before and after the first intervention)
  To estimate the level of depression among adults, this scale has 13 items with a 4-points Likert scale (0 to 3). The score ranges from 0 to 39, a higher score means a higher level of depression.
Beck Depression Scale | Month 2 (a week after the second intervention)
  To estimate the level of depression among adults, this scale has 13 items with a 4-points Likert scale (0 to 3). The score ranges from 0 to 39, a higher score means a higher level of depression.
Beck Depression Scale | Month 3
  To estimate the level of depression among adults, this scale has 13 items with a 4-points Likert scale (0 to 3). The score ranges from 0 to 39, a higher score means a higher level of depression.
Fat/lean mass ratio | Month 1 (Between 1 day and a week before and after the first intervention)
  The bio-electrical impedance analysis measurements will include total body fat mass (FM in kg), and total body lean mass (LM in kg). Then the fat/lean mass (F/L) ratio will be calculated.
Fat/lean mass ratio | Month 2 (a week after the second intervention)
  The bio-electrical impedance analysis measurements will include total body fat mass (FM in kg), and total body lean mass (LM in kg). Then the fat/lean mass (F/L) ratio will be calculated.
Fat/lean mass ratio | Month 3
  The bio-electrical impedance analysis measurements will include total body fat mass (FM in kg), and total body lean mass (LM in kg). Then the fat/lean mass (F/L) ratio will be calculated.
Client satisfaction questionnaire | Month 1 (Between 1 day and a week before and after the first intervention)
  This survey assesses the patient's satisfaction level of the intervention. Eight items with a 4-points Likert scale (1 to 4) allow to obtain a score between 8 and 32. A higher score means a better satisfaction level.
Client satisfaction questionnaire | Month 2 (a week after the second intervention)
  This survey assesses the patient's satisfaction level of the intervention. Eight items with a 4-points Likert scale (1 to 4) allow to obtain a score between 8 and 32. A higher score means a better satisfaction level.
Client satisfaction questionnaire | Month 3
  This survey assesses the patient's satisfaction level of the intervention. Eight items with a 4-points Likert scale (1 to 4) allow to obtain a score between 8 and 32. A higher score means a better satisfaction level.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Magnon V, Dutheil F, Tauveron I, Mille J, Baker JS, Brusseau V, Silvert L, Izaute M, Vallet GT. Does an increase in physiological indexes predict better cognitive performance: the PhyCog randomised cross-over protocol in type 2 diabetes. BMJ Open. 2022 Jul 1;12(7):e060057. doi: 10.1136/bmjopen-2021-060057. PMID 35777867